CLINICAL TRIAL: NCT06995677
Title: A Phase 2 Multicenter, Open-Label Study Evaluating the Efficacy and Safety of TYRA-300 in Participants With FGFR3 Altered Low Grade, Intermediate Risk Non-Muscle Invasive Bladder Cancer (SURF302)
Brief Title: Efficacy and Safety of TYRA-300 in Participants With FGFR3 Altered Low Grade, Intermediate Risk Non-Muscle Invasive Bladder Cancer
Acronym: SURF302
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYR300-202
Record Dates: First submitted 2025-04-25; First posted 2025-05-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Low-grade NMIBC; FGFR Gene Amplification; FGFR Gene Alterations; FGFR3 Gene Alteration; FGFR3 Gene Mutation; FGFR3 Gene Fusions
Keywords: FGFR3 gene alterations; FGFR3 gene mutations; FGFR3 gene fusions; FGFR3; Non-Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort A will test a TYRA-300 dose of 60mg QD. In addition, Dose Cohort B will test, in parallel, a slightly reduced dose of TYRA-300 50 mg QD. Dose Cohort C of TYRA-300 will only open if another dose needs to be explored based on the safety and efficacy results from Cohorts A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Cohort A (DCA) (Experimental): TYRA-300 monotherapy in Participants with FGFR3 Altered Low Grade, Intermediate Risk Non-Muscle Invasive Bladder Cancer
  Interventions: Drug: TYRA-300 60mg
- Dose Cohort B (DCB) (Experimental): TYRA-300 monotherapy in Participants with FGFR3 Altered Low Grade, Intermediate Risk Non-Muscle Invasive Bladder Cancer
  Interventions: Drug: TYRA-300 50mg
- Possible Dose Cohort C (DCC) (Experimental): To Be Determined- TYRA-300 monotherapy in Participants with FGFR3 Altered Low Grade, Intermediate Risk Non-Muscle Invasive Bladder Cancer
  Interventions: Drug: TYRA-300 Dose TBD

INTERVENTIONS:
Drug: TYRA-300 60mg — Self-administered 60mg dose Oral tablet(s) given daily
  Arms: Dose Cohort A (DCA)
Drug: TYRA-300 50mg — Self-administered 50mg dose Oral tablet(s) given daily
  Arms: Dose Cohort B (DCB)
Drug: TYRA-300 Dose TBD — To Be Determined Dose: Self-administered Oral tablet(s) given daily
  Arms: Possible Dose Cohort C (DCC)

SUMMARY:
Phase 2 Study of TYRA-300 in FGFR3 Altered Low Grade, Intermediate Risk NMIBC

DETAILED DESCRIPTION:
A Phase 2 Multicenter, Open-Label Study Evaluating the Efficacy and Safety of TYRA-300 in Participants with FGFR3 Altered Low Grade, Intermediate Risk Non-Muscle Invasive Bladder Cancer

ELIGIBILITY:
Inclusion Criteria:

* Participants age 18 and over of informed consent and willing and able to comply with all requires study procedures
* Able to understand and given written informed consent
* Participants with histologically confirmed low-grade NMIBC within 6 weeks prior to randomization with prior diagnostic biopsy/TURBT to confirm stage and grade and with at least 3 mm and no more than 12 mm total (1/2 a resectoscope loop to 2 loops, refer to Section 8.1.5) residual visible tumor as a marker lesion(s) left behind:

  1. Ta low grade
  2. T1 low grade
* Participants must have intermediate risk NMIBC, defined as having any of the following characteristics (AUA Guidelines, 2024)

  1. Recurrence within 1 year, LG Ta
  2. Solitary LG Ta >3cm
  3. LG Ta, multifocal
  4. LG T1
* Documented activating FGFR3 mutation or fusion (Appendix 4)
* Have undergone bladder mapping and identification of visible marker lesion(s) within 6 weeks prior to randomization (refer to Inclusion Criterion #3)
* No evidence of urothelial carcinoma of the upper urinary tract (confirmed by imaging) or prostatic urethra within 6 months of randomization
* No prior BCG administration within 1 year of date of consent.
* No intravesical chemotherapy within 8 weeks prior to C1D1.
* ECOG 0-1
* Pathology consistent with pure urothelial carcinoma; if mixed histology, ensure that at least 80% of the sample is urothelial
* Adequate bone marrow, liver, and renal function:

  b. Bone marrow function: i. Absolute neutrophil count (ANC) > or = 1,500/mm3 ii. Platelet count > or = 75,000/mm3 iii. /hemoglobin > or = 10.0 g/dL e. Liver function: i.Total bilirubin < or = ULN ii. Alanine aminotransferase (ALT) < or = ULN iii. Aspartate aminotransferase (AST) < or = ULN f. Renal function: i. estimated glomerular filtration rate >60 mL/min calculated using the modification of diet in renal disease equation or CKD-EPI formula ii. Serum Phosphate level < or = ULN prior to starting treatment g. Coagulation i. International normalized ratio (INR) < or = 1.5 x ULN
* Ability to swallow tablets
* Participants (male and female) of child-bearing potential (including females who are post-menopausal for less than 1 year) must be willing to practice effective contraception while on treatment and be willing and able to continue contraception for 3 months (males) and 6 months (females) after the last dose of study treatment. Potential male participants should consider the potential impact of TYRA-300 on their ability to father a child and discuss options with the site study staff.
* Potential participants who are positive for human immunodeficiency virus (HIV) must have a viral load below the limits of detection and on stable antiretroviral therapy for at least 3 months prior to C1D1. NOTE: some of the compounds in antiretroviral therapy may be on the prohibited medications list. Allowances will be made to ensure the participant's HIV treatment continues uninterrupted following a discussion with the Sponsor's medical monitor. A discussion of the impact of the antiretroviral therapy on TYRA- 300 needs to be discussed with the potential participant prior to C1D1.
* Potential participants with chronic hepatitis B virus (HBV) infection with active disease should be on a suppressive antiviral therapy prior to C1D1.
* Potential participants patients with a history of hepatitis C virus (HCV) infection should have completed curative antiviral treatment and must have a HCV viral load below the limit of quantification.
* Potential participants with a history of HCV infection and on current treatment must have a HCV viral load below the limit of quantification

Exclusion Criteria:

* Presence of tumor in ureter or prostatic urethra:
* Current or previous history of muscle invasive bladder cancer
* Current or previous history of lymph node positive and/or metastatic bladder cancer
* Evidence of pure squamous cell carcinoma, pure adenocarcinoma or pure undifferentiated carcinoma of the bladder
* Currently receiving systemic cancer therapy (cytotoxic, immunotherapy, targeted)
* Currently receiving treatment with a prohibited therapy (refer to Section 6.7.1)
* Current or prior history of pelvic external beam radiotherapy
* Current or history of receiving a prior FGFR inhibitor
* Systemic immunotherapy within 6 months prior to randomization
* Treatment with an investigational agent within 30 days or 5 half-lives from randomization, whichever is shorter; compounds with an unknown half-life will default to the 30 days.
* Prior treatment with an intravesical agent within 8 weeks prior to C1D1
* Current ongoing toxicity from previous therapy
* Had major surgery within 4 weeks prior to C1D1
* Any reason that in the view of the investigator, would substantially impair the ability of the participant to comply with study procedures and/or risk to the participant (i.e., uncontrolled diabetes)
* Females who are pregnant, breastfeeding or planning to become pregnant within 6 months after the last dose of TYRA-300 and males who plan to father a child while enrolled in this study or within 3 months after the last dose of TYRA-300
* Has impaired wound healing capacity
* Serum phosphate levels above the upper limit of normal during screening
* Any ocular condition likely to increase the risk of eye toxicity
* Current evidence of central serous retinopathy or retinal pigmented epithelial detachment of any grade at time of baseline examination.
* History of or current uncontrolled cardiovascular disease
* Gastrointestinal disorders that will affect oral administration or absorption of TYRA-300
* Known history of HIV infection, or active hepatitis B or C
* History of a second primary malignancy within 3 years of signing ICF, except for nonmelanoma skin cancer and cured and active surveillance malignancies (i.e., prostate, breast) .
* Known allergy to TYRA-300 or any excipients of the formulated product
* Participants taking strong inhibitors and/or inducers of CYP3A4 enzyme
* History of prolonged QT syndrome or baseline heart rate-corrected QT interval using Fridericia formula (QTcF) interval >470 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of TYRA-300 in LG IR-NMIBC participants | at 3 months
  Complete response (CR) rate

SECONDARY OUTCOMES:
Duration of response (responders only) | time from initial response to confirmed recurrence of disease or death, up to 24 months
Time to recurrence (responders only) | time from start of response to confirmed recurrence of disease, up to 24 months
Recurrence-free survival rate (responders only) | at 12 months and 24 months
Progression-free survival (all participants) | time from randomization to the progression of disease or death from any cause, whichever occurs first, up to 24 months
Incidence and severity of adverse events | Up to 2 years
To assess the safety and tolerability of TYRA-300 in LG IR-NMIBC participants | From initiation of treatment to 2 years
  Assessed by adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Doug Warner, MD, Study Chair — Tyra Biosciences, Inc
Locations (16):
- United States (12):
  - Urology Centers of Alabama, Homewood, Alabama
  - Tri Valley Urology - Murrieta, Murrieta, California
  - Genesis Research, San Diego, California
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - The Bronx Veterans Medical Research Foundation, Inc., The Bronx, New York
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Lowcounty Urology Clinics, P.A., North Charleston, South Carolina
  - Urology Associates PC, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Istituti Fisioterapici Ospitalieri (IFO), Rome, Italy, Italy
- Spain (3):
  - Centro Médico Teknon, Barcelona, Spain
  - Hospital Clínico San Carlos, Madrid, Spain
  - Hospital Universitario 12 de Oc, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No